CLINICAL TRIAL: NCT01912716
Title: Rectal Indomethacin in the Prevention of Post-ERCP Pancreatitis in High Risk Patients: Searching for the Optimal Dose. A Prospective, Randomized Trial
Brief Title: Rectal Indomethacin in the Prevention of Post-ERCP Pancreatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American College of Gastroenterology (Other); University of Michigan (Other); University of Texas (Other); Wake Forest University Health Sciences (Other); Medical University of South Carolina (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Evan Fogel, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEP INDO 2013; ACG-CR-002-2013 (Other Grant/Funding Number: American College of Gastroenterology)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Post-ERCP Pancreatitis
Keywords: pancreatitis; ERCP
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high-dose indomethacin (Experimental): 200mg rectal indomethacin
  Interventions: Drug: high dose indomethacin
- standard dose indomethacin (Active Comparator): 100mg rectal indomethacin
  Interventions: Drug: standard dose indomethacin

INTERVENTIONS:
Drug: high dose indomethacin — patients randomized to this intervention receive 200mg indomethacin
  Other Names: Indocin
  Arms: high-dose indomethacin
Drug: standard dose indomethacin — patients randomized to this intervention receive 100mg indomethacin
  Other Names: Indocin
  Arms: standard dose indomethacin

SUMMARY:
It is now established that indomethacin, a non-steroidal anti-inflammatory drug, at a dose of 100 mg, is effective in reducing the frequency and severity of pancreatitis (inflammation of the pancreas) after endoscopic retrograde cholangiopancreatography (ERCP) in high risk patients. However, the optimal dose required is not known. The purpose of this study is to determine whether a dose of 200 mg, administered as rectal suppositories, is more effective than the standard dose of 100 mg. An ERCP procedure is a scope procedure where a lighted tube with a camera is passed down the patient's throat and allows for evaluation of the bile duct and/or pancreatic duct. The most common side effect of this procedure is post-ERCP pancreatitis, or swelling of the pancreas. Some patients are at higher risk for this complication than others. Our hypothesis is to compare the efficacy of these two dose regimens (100 mg vs 200 mg) of prophylactic rectally-administered indomethacin on the frequency and severity of post-ERCP pancreatitis in high-risk patients.

DETAILED DESCRIPTION:
After obtaining informed consent, subjects will undergo ERCP per clinical protocol. All procedure-related clinical decisions and interventions will be dictated by the performing physician as he or she sees fit. At the end of the procedure, it will be determined by the endoscopist and research coordinator whether the patient meets inclusion criteria. If inclusion criteria are met, subjects will be randomized by concealed allocation to receive either 100mg or 150mg indomethacin, in the form of two or three 50mg rectal suppositories. Those patients who are randomized to receive the 100mg dose will receive an additional glycerin suppository. Four hours later, those patients who were randomized to the high-dose group will then receive an additional 50mg suppository while in the recovery area. At this same time point, subjects who were randomized to the standard-dose group, will receive a glycerin suppository in the recovery area. All participating patients will receive a total of 4 suppositories.

ELIGIBILITY:
Inclusion Criteria:

Included patients are those undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) and have:

one of the following:

1. Clinical suspicion of sphincter of Oddi dysfunction (SOD; type I or II)
2. History of post-ERCP pancreatitis (at least one episode)
3. Pancreatic sphincterotomy
4. Pre-cut (access) sphincterotomy
5. greater than 8 cannulation attempts of any sphincter
6. Pneumatic dilation of intact biliary sphincter
7. Ampullectomy 8.) Assessment for post-sphincterotomy stenosis

OR at least 2 of the following:

1. Age less than 50 years old and female gender
2. History of recurrent pancreatitis (at least 2 episodes)
3. greater than or equal to to 3 pancreatic injections, with at least 1 injection to tail
4. Pancreatic acinarization (excluding ventral pancreas of pancreas divisum)
5. Pancreatic brush cytology -

Exclusion Criteria:

1. Unwillingness or inability to consent for the study
2. Age less than 18 years
3. Intrauterine pregnancy
4. Breastfeeding mother
5. Standard contraindications to ERCP
6. Allergy/hypersensitivity to aspirin or Nonsteroidal Anti-Inflammatory Drugs (NSAIDs)
7. Received NSAIDs in prior 7 days (aspirin 325mg or less ok)
8. Renal failure (serum creatinine greater than 1.4)
9. Active or recurrent (within 4 weeks) gastrointestinal hemorrhage
10. Acute pancreatitis (lipase peak) within 72 hours
11. Known chronic calcific pancreatitis
12. Pancreatic head mass
13. Procedure performed on major papilla/ventral pancreatic duct in patient with pancreas divisum (dorsal duct not attempted on injected)
14. ERCP for biliary stent removal or exchange without anticipated pancreatogram
15. Subject with prior biliary sphincterotomy now scheduled for repeat biliary therapy without anticipated pancreatogram
16. Anticipated inability to follow protocol
17. Known active cardiovascular or cerebrovascular disease -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1037 (Actual)
Dates: Start 2013-07; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Fogel, MD, MSc, Principal Investigator — Indiana University Health
Locations (6):
- United States (6):
  - Indiana University Health, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Aurora St. Lukes' Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fogel EL, Lehman GA, Tarnasky P, Cote GA, Schmidt SE, Waljee AK, Higgins PDR, Watkins JL, Sherman S, Kwon RSY, Elta GH, Easler JJ, Pleskow DK, Scheiman JM, El Hajj II, Guda NM, Gromski MA, McHenry L Jr, Arol S, Korsnes S, Suarez AL, Spitzer R, Miller M, Hofbauer M, Elmunzer BJ; US Cooperative for Outcomes Research in Endoscopy (USCORE). Rectal indometacin dose escalation for prevention of pancreatitis after endoscopic retrograde cholangiopancreatography in high-risk patients: a double-blind, randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Feb;5(2):132-141. doi: 10.1016/S2468-1253(19)30337-1. Epub 2019 Nov 25. PMID 31780277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between July 2013 - March 2018, either from the ERCP (Endoscopic Retrograde Cholangiopancreatography) outpatient clinic or Peri-Operative Care Unit immediately prior to ERCP.
Groups:
- High-dose Indomethacin: 200mg rectal indomethacin
  high dose indomethacin
- Standard Dose Indomethacin: 100mg rectal indomethacin
  standard dose
Period: Overall Study
Arm/Group | High-dose Indomethacin | Standard Dose Indomethacin
Started | 522 (receipt of 1st dose of indomethacin) | 515
Receipt of 2nd Dose | 511 | 503
5-day Follow-up | 522 | 515
3-day Follow-up | 521 | 513
Completed | 522 | 515
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Dose Group: Participants randomized to this group receive 100 mg indomethacin
- High Dose Group: Participants randomized to this group receive 200 mg indomethacin
- Total: Total of all reporting groups
Arm/Group | Standard Dose Group | High Dose Group | Total
Number analyzed (Participants) | 515 | 522 | 1037
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (15.2) | 50.4 (15) | 49.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 392 | 421 | 813
  Male | 123 | 101 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 35
  Not Hispanic or Latino | 493 | 507 | 1000
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 12 | 28
  White | 485 | 501 | 986
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 9 | 4 | 13
BMI [Geometric Mean (Standard Deviation); unit: kg/m^2] | 28.6 (7.0) | 29.2 (7.6) | 28.9 (7.3)
Obese [Count of Participants; unit: Participants] — BMI greater than or equal to 30
  Participants | 193 | 198 | 391
Clinical Suspicion of SOD (sphincter of Oddi dysfunction) [Count of Participants; unit: Participants] | 319 | 331 | 650
History of post-ERCP pancreatitis [Count of Participants; unit: Participants] | 77 | 100 | 177
History of recurrent pancreatitis [Count of Participants; unit: Participants] | 202 | 210 | 412
Difficult Cannulation [Count of Participants; unit: Participants] — greater than 8 attempts at cannulation of desired duct
  Participants | 148 | 146 | 294
Precut sphincterotomy [Count of Participants; unit: Participants] | 71 | 46 | 117
Double-wire cannulation technique [Count of Participants; unit: Participants] | 18 | 18 | 36
Pancreatography (patients) [Count of Participants; unit: Participants] | 446 | 433 | 879
Number of pancreatic duct injections [Geometric Mean (Standard Deviation); unit: injections] | 2.12 (1.63) | 1.96 (1.66) | 2.04 (1.64)
Therapeutic pancreatic sphincterotomy [Count of Participants; unit: Participants] | 245 | 231 | 476
Placement of pancreatic stent [Count of Participants; unit: Participants] | 400 | 393 | 793
Ampullectomy [Count of Participants; unit: Participants] | 30 | 32 | 62
Biliary sphincterotomy [Count of Participants; unit: Participants] | 302 | 290 | 592
Trainee involvement [Count of Participants; unit: Participants] | 84 | 68 | 152

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Post-ERCP Pancreatitis
Description: Assessment of whether patients developed post-ERCP pancreatitis, defined as a new onset of pain (or worsening of existing pain) in the upper abdomen, an elevation in pancreatic enzymes of at least three times the upper limit of the normal range 24 hours after the procedure, and hospitalization for at least two nights.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Standard 100mg Dose: patients receiving 100mg indomethacin
- High Dose 200 mg: patients receiving 200mg indomethacin
Arm/Group | Standard 100mg Dose | High Dose 200 mg
Number analyzed (Participants) | 515 | 522
Participants | 76 | 65

2. Secondary Outcome: Number of Participants With Moderate or Severe Post-ERCP Pancreatitis
Description: Assessment of whether patients developed either moderate or severe post-ERCP pancreatitis, defined according to established consensus criteria (Cotton et al., Gastrointestinal Endoscopy 1991;37:383-93). Severity of post-ERCP pancreatitis is partly defined according to length of stay. Moderate pancreatitis is defined as a 4-10 day hospitalization. Severe post-ERCP pancreatitis is defined as a hospitalization of greater than 10 days post-ERCP, or development of a complication (eg. pseudocyst or necrosis), or need for intervention (drainage or surgery).
Time Frame: 30 days
Population: development of moderate or severe post-ERCP pancreatitis
Measure: Count of Participants; unit: Participants
Groups:
- Standard Dose 100 mg: patients receiving 100mg indomethacin
- High Dose 200mg: patients receiving 200mg indomethacin
Arm/Group | Standard Dose 100 mg | High Dose 200mg
Number analyzed (Participants) | 515 | 522
Participants | 28 | 28

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the length of the study, i.e. 5 years. Patients were recruited from July 2013 until March 2018. Following recruitment of the last patient (i.e. #1037), follow-up for an additional 30-day period was undertaken to capture severity of pancreatitis (should it occur) and delayed adverse events.
Description: In this study, there was no difference in definition of adverse events or serious adverse events, as other [not including serious] adverse events were not monitored/assessed. All patients provided contact information (home phone, cell phone, personal e-mail address) at study entry, and patients were then contacted at 5 and 30 days to assess for these adverse events, as noted in the study protocol.
Groups:
- Standard-dose Indomethacin: 100mg rectal indomethacin
  standard dose indomethacin
- High-dose Indomethacin: 200mg rectal indomethacin
  high-dose dose
Arm/Group | Standard-dose Indomethacin | High-dose Indomethacin
All-Cause Mortality (participants affected / at risk) | 0/515 | 0/522
Serious Adverse Events (participants affected / at risk) | 83/515 | 77/522
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-dose Indomethacin (N=515) | High-dose Indomethacin (N=522)
pancreatitis (Gastrointestinal disorders) | 76 (76) | 65 (65) — requiring hospitalization. Definition of post-ERCP pancreatitis was according to established consensus criteria (Cotton et al., Gastrointestinal Endoscopy 1991;37:383-93).
bleeding (Gastrointestinal disorders) | 6 (6) | 8 (8) — as per consensus criteria (as noted for pancreatitis definition)
renal failure (Renal and urinary disorders) | 0 (0) | 3 (3) — increase in baseline serum creatinine, to greater than 1.4
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
allergy (Immune system disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study took place at 6 tertiary medical centers in the United States. However, approximately 3/4 of patients were enrolled from a single site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT01912716/Prot_SAP_001.pdf